CLINICAL TRIAL: NCT07013253
Title: Burnout Syndrome Among Anesthesiology Residents in Turkey: A Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Leman Gökçenur Aydın, Medical Doctor, Uludag University
Other Study IDs: 2025-2/13
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Burnout, Professional; Burnout, Psychological
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burnout syndrome is a condition in which an individual experiences loss of self-esteem, chronic fatigue, feelings of helplessness, and hopelessness in their professional work life and human relationships. This study aims to evaluate the prevalence of burnout syndrome among anesthesiology residents working in Turkey, analyze the potential causes and adverse consequences of this syndrome's increase, and provide recommendations for its reduction.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate by completing the online survey form
* Proficient in the Turkish language
* Anesthesiology and Reanimation residents currently practicing in the Republic of Turkey

Exclusion Criteria:

• Participants who do not provide consent to share the requested information in the survey form

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anesthesiology and Reanimation residents currently practicing in the Republic of Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Burnout Syndrome as measured by the Maslach Burnout Inventory | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Selcan Akesen, Assc Prof, Study Chair — Uludağ Üniversitesi